CLINICAL TRIAL: NCT07340515
Title: A Prospective, Randomized, Open-Label, Multicenter Phase III Clinical Study Comparing Intensity-Modulated Proton Therapy and Intensity-Modulated Photon Radiotherapy in Locally Advanced Nasopharyngeal Carcinoma
Brief Title: Proton vs Photon IMRT in Locally Advanced Nasopharyngeal Carcinoma: A Phase III Trial
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Man Hu (Other)
Collaborators: Shandong Cancer Hospital and Institute (Other)
Responsible Party: Sponsor-Investigator, Man Hu, Chief Physician, Shandong Cancer Hospital and Institute
Organization: Shandong Cancer Hospital and Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025XH13
Record Dates: First submitted 2025-12-09; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-11

CONDITIONS: Nasopharyngeal Carcinoma (NPC)
Keywords: Proton Therapy; IMPT; Intensity-Modulated Proton Therapy; Nasopharyngeal Carcinoma; Chemoradiotherapy
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Radiotherapy, Intensity-Modulated; Cisplatin; toripalimab

STUDY DESIGN:
Intervention Model Description: Participants are randomized in a 1:1 ratio to receive intensity-modulated proton therapy (IMPT) or intensity-modulated photon radiotherapy (IMRT) using a parallel-group design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IMPT Arm (Experimental): Participants assigned to this arm receive intensity-modulated proton therapy (IMPT). Radiotherapy is delivered according to the protocol-defined dose and fractionation schedule, using the same target delineation and prescription principles as IMRT, with dose converted to Gy(RBE) for proton therapy. IMPT treatment is administered concurrently with cisplatin-based chemotherapy and toripalimab as specified in the study protocol.
  Interventions: Radiation: Intensity-Modulated Proton Therapy (IMPT); Drug: Cisplatin; Biological: Toripalimab
- IMRT Arm (Active Comparator): Participants assigned to this arm receive intensity-modulated photon radiotherapy (IMRT) according to the protocol-defined dose and fractionation schedule. Radiotherapy is delivered to the primary tumor and involved lymph nodes following the target delineation and prescription principles specified in the study protocol. IMRT is administered concurrently with cisplatin-based chemotherapy and toripalimab, consistent with the protocol.
  Interventions: Radiation: Intensity-Modulated Radiation Therapy (IMRT); Drug: Cisplatin; Biological: Toripalimab

INTERVENTIONS:
Radiation: Intensity-Modulated Proton Therapy (IMPT) — Participants assigned to this arm receive intensity-modulated proton therapy (IMPT) according to the protocol-defined dose and fractionation schedule. Radiotherapy is delivered using the same target delineation and prescription principles as IMRT, with dose converted to Gy(RBE) for proton therapy. IMPT is administered concurrently with cisplatin-based chemotherapy and toripalimab as specified in the study protocol.
  Arms: IMPT Arm
Radiation: Intensity-Modulated Radiation Therapy (IMRT) — Participants assigned to this arm receive intensity-modulated radiation therapy (IMRT) according to the protocol-defined dose and fractionation schedule. Radiotherapy is delivered to the primary tumor and involved lymph nodes following the target delineation and prescription principles specified in the study protocol. IMRT is administered concurrently with cisplatin-based chemotherapy and toripalimab, consistent with the protocol.
  Arms: IMRT Arm
Drug: Cisplatin — Cisplatin is administered during induction chemotherapy and concurrent chemoradiotherapy as specified in the protocol: 80 mg/m² IV on Day 1 every 21 days for 3 cycles during induction (GP regimen), and 100 mg/m² IV on Day 1 and Day 22 for 2 cycles during concurrent chemoradiotherapy.
Biological: Toripalimab — Toripalimab 240 mg is administered every 3 weeks during induction, concurrent chemoradiotherapy, and maintenance therapy for a total of 12 cycles unless disease progression or unacceptable toxicity occurs.

SUMMARY:
This multicenter, open-label, randomized Phase III trial evaluates intensity-modulated proton therapy (IMPT) versus intensity-modulated photon radiotherapy (IMRT) in patients with newly diagnosed, high-risk, locoregionally advanced nasopharyngeal carcinoma.

All patients receive induction chemotherapy followed by concurrent chemoradiotherapy combined with immunotherapy and are randomized 1:1 to IMPT or IMRT during the concurrent treatment phase.

The primary endpoints are the incidence of grade ≥3 acute treatment-related toxicities and the 3-year progression-free survival (PFS) rate. Secondary endpoints include overall survival, locoregional relapse-free survival, distant metastasis-free survival, objective response rate, late toxicities, and quality of life.

DETAILED DESCRIPTION:
This is a multicenter, open-label, randomized Phase III clinical trial designed to compare the safety and efficacy of intensity-modulated proton therapy (IMPT) versus intensity-modulated photon radiotherapy (IMRT) in patients with newly diagnosed, high-risk, locoregionally advanced nasopharyngeal carcinoma.

Eligible patients are adults aged 18 to 70 years with histologically confirmed non-keratinizing nasopharyngeal carcinoma (WHO type II or III) and clinical stage T4 or N3 disease without distant metastasis (M0), according to the AJCC staging system.

All enrolled patients will receive three cycles of induction chemotherapy consisting of gemcitabine plus cisplatin. This will be followed by concurrent chemoradiotherapy combined with immunotherapy. During the concurrent treatment phase, patients will be randomized in a 1:1 ratio to receive either IMPT or IMRT, delivered according to protocol-defined target delineation, dose prescription, and fractionation schedules.

The first primary endpoint is the incidence of grade ≥3 acute treatment-related toxicities, defined as treatment-related adverse events of grade 3 or higher occurring from the initiation of radiotherapy to 90 days after completion of radiotherapy. Toxicities will be graded according to CTCAE version 5.0 and RTOG criteria. Ototoxicity, including hearing loss or tinnitus, will be further evaluated using the ASHA (1994) significant change criteria for pure-tone audiometry.The second primary endpoint is the 3-year progression-free survival (PFS) rate, defined as the proportion of patients who remain alive without documented disease progression within 3 years after randomization. Disease progression is defined as locoregional recurrence, distant metastasis, or death from any cause, whichever occurs first.

Secondary endpoints include overall survival (OS), defined as the time from randomization to death from any cause; locoregional relapse-free survival (LRRFS), defined as the time from enrollment to the first occurrence of locoregional recurrence; distant metastasis-free survival (DMFS), defined as the time from randomization to the first occurrence of distant metastasis; objective response rate (ORR), defined as the proportion of patients achieving complete response (CR) or partial response (PR), assessed at 2 weeks after completion of induction chemotherapy and at 3 months after completion of radiotherapy; incidence of grade <3 acute toxicities; and incidence and severity of late treatment-related toxicities assessed according to CTCAE version 5.0.Quality of life will be evaluated using the European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire Core 30 (QLQ-C30, version 3.0) and the Head and Neck Cancer-specific module QLQ-H&N35 (version 1.0), administered at baseline, at the end of treatment, and during follow-up visits.

The trial aims to determine whether IMPT can reduce treatment-related toxicities while maintaining or improving disease control and survival outcomes compared with IMRT.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 70 years
* Histologically confirmed nasopharyngeal carcinoma (WHO type II or III)
* High-risk locoregionally advanced disease defined as clinical stage T4 or N3, M0, according to the AJCC staging system
* No prior anti-tumor therapy for nasopharyngeal carcinoma, including radiotherapy, chemotherapy, targeted therapy, or immunotherapy
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Adequate organ function as defined in the study protocol
* Eligible to receive induction chemotherapy followed by concurrent chemoradiotherapy combined with immunotherapy as specified in the protocol
* Ability to understand and willingness to sign written informed consent

Exclusion Criteria:

* Evidence of distant metastasis (M1 disease)
* Prior radiotherapy, chemotherapy, targeted therapy, or immunotherapy for nasopharyngeal carcinoma
* Active autoimmune disease requiring systemic therapy
* Uncontrolled infection or severe comorbidities that may affect treatment tolerance
* Pregnancy or breastfeeding
* Known allergy, hypersensitivity, or contraindication to study medications as defined in the protocol
* Any other condition that, in the investigator's judgment, makes the patient unsuitable for participation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2031-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-related grade ≥3 acute toxicities | From the start of radiotherapy to 90 days after completion of radiotherapy
  The proportion of patients who experience treatment-related grade ≥3 acute toxicities, defined as adverse events occurring from the start of radiotherapy to 90 days after completion of radiotherapy, assessed according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 and Radiation Therapy Oncology Group (RTOG) criteria. Ototoxicity (hearing loss or tinnitus), if present, will additionally be evaluated using the American Speech-Language-Hearing Association (ASHA, 1994) significant change criteria.
3-year Progression-Free Survival (PFS) Rate | 3 years
  Defined as the proportion of participants who remain alive and progression-free at 3 years after randomization, with progression-free survival events defined as disease progression or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Overall Survival (OS) | 3 years
  Defined as the time interval from randomization to death due to any cause.
Locoregional Recurrence-Free Survival (LRRFS) | 3 years
  Defined as the time from randomization to the date of first locoregional relapse.
Distant Metastasis-Free Survival (DMFS) | 3 years
  Defined as the time interval from randomization to the date of first distant metastasis.
Objective Response Rate (ORR) | 2 weeks after induction chemotherapy and 3 months after completion of radiotherapy
  Defined as the proportion of participants who achieve a complete response (CR) or partial response (PR). Tumor response will be evaluated 2 weeks after completion of induction chemotherapy and 3 months after completion of radiotherapy.
Incidence of Grade <3 Acute Treatment-Related Toxicities | From the start of radiotherapy to 90 days after completion of radiotherapy
  The proportion of participants who experience treatment-related acute adverse events of grade <3. Acute toxicities include anemia, leukopenia, neutropenia, nausea, oral mucositis, anorexia, xerostomia, dermatitis/skin inflammation, fatigue, vomiting, weight loss, and hearing loss.
Incidence of treatment-related late toxicities | From 90 days after completion of radiotherapy up to 3 years
  The proportion of patients who experience treatment-related late toxicities occurring more than 90 days after completion of radiotherapy, assessed according to CTCAE version 5.0 and RTOG late radiation morbidity scoring criteria.
Score of quality of life according to the EORTC Quality of Life Questionnaire (QLQ)-C30 (V3.0) | Up to 3 years
  Quality of life will be assessed using the European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire Core 30 (QLQ-C30, version 3.0). The QLQ-C30 consists of multi-item functional scales, symptom scales, and a global health status/quality of life scale. All scale scores range from 0 to 100. For functional scales and global health status, higher scores indicate better functioning or quality of life, whereas for symptom scales, higher scores indicate worse symptom burden.Assessments will be performed before treatment, during treatment, and after completion of treatment.
Score of quality of life according to the EORTC Quality of Life Questionnaire Head and Neck Module (QLQ-H&N35) | Up to 3 years
  Head and neck cancer-specific quality of life will be evaluated using the European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire Head and Neck Module (QLQ-H&N35).The QLQ-H&N35 is a disease-specific module designed to assess symptoms and functional impairments related to head and neck cancer and its treatment. All scale scores range from 0 to 100, with higher scores indicating worse symptom severity or functional impairment.Assessments will be conducted before treatment, during treatment, and after completion of treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Shandong Cancer Hospital and Institute, Shandong First Medical University and Shandong Academy of Medical Sciences, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No